CLINICAL TRIAL: NCT00316771
Title: A Randomized, Double-blind, Placebo-controlled, Study to Determine the Efficacy and Safety of 5 Dose Regimens of RO4402257 in Patients With Active Rheumatoid Arthritis (RA) on Stable Methotrexate (MTX) Therapy.
Brief Title: A Study of P38 Inhibitor (4) in Patients With Active Rheumatoid Arthritis (RA) on Stable Methotrexate Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA18439
Record Dates: First submitted 2006-04-20; First posted 2006-04-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- P38 Inhibitor (4) 150mg (Experimental)
  Interventions: Drug: P38 Inhibitor (4) 150mg
- P38 Inhibitor (4) 25mg (Experimental)
  Interventions: Drug: P38 Inhibitor (4) 25mg
- P38 Inhibitor (4) 300mg (Experimental)
  Interventions: Drug: P38 Inhibitor (4) 300mg
- P38 Inhibitor (4) 50mg (Experimental)
  Interventions: Drug: P38 Inhibitor (4) 50mg
- P38 Inhibitor (4) 75mg (Experimental)
  Interventions: Drug: P38 Inhibitor (4) 75mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: P38 Inhibitor (4) 150mg — 150mg po qd
  Arms: P38 Inhibitor (4) 150mg
Drug: P38 Inhibitor (4) 25mg — 25mg po bid
  Arms: P38 Inhibitor (4) 25mg
Drug: P38 Inhibitor (4) 300mg — 300mg po qd
  Arms: P38 Inhibitor (4) 300mg
Drug: P38 Inhibitor (4) 50mg — 50mg po qd
  Arms: P38 Inhibitor (4) 50mg
Drug: P38 Inhibitor (4) 75mg — 75mg po bid
  Arms: P38 Inhibitor (4) 75mg
Drug: Placebo — po bid
  Arms: Placebo

SUMMARY:
This 6 arm study will evaluate the efficacy and safety of different doses of P38 Inhibitor (4) in patients with RA currently having an inadequate clinical response to methotrexate. Patients will be randomized to receive P38 Inhibitor (4) (50,150 or 300 qd po,and 25 or 75 bid po) or placebo, and will remain on the stable dose of methotrexate. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* active rheumatoid arthritis;
* current inadequate clinical response to methotrexate.

Exclusion Criteria:

* receiving any other disease-modifying anti-rheumatic drug, with the exception of hydroxychloroquine or chloroquine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2005-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ACR 20 response | Week 12

SECONDARY OUTCOMES:
Percentage of patients with ACR 50/70 response | Week 12
Change in ACR core set, DAS 28, HAQ disability index, SF-36, withdrawals, AEs, lab parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (103):
- United States (45):
  - Birmingham, Alabama
  - Paradise Valley, Arizona
  - Tucson, Arizona
  - Escondido, California
  - Fair Oaks, California
  - Loma Linda, California
  - Riverside, California
  - Upland, California
  - Gainesville, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Sarasota, Florida
  - Tamarac, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Nampa, Idaho
  - Munster, Indiana
  - South Bend, Indiana
  - Wichita, Kansas
  - Worcester, Massachusetts
  - Traverse City, Michigan
  - Omaha, Nebraska
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - New Hartford, New York
  - Rochester, New York
  - Belmont, North Carolina
  - North Fargo, North Dakota
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Camp Hill, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Sioux Falls, South Dakota
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Amarillo, Texas
  - Bryan, Texas
  - Carrollton, Texas
  - Lubbock, Texas
  - Norfolk, Virginia
  - Everett, Washington
  - Seattle, Washington
  - Monroe, Wisconsin
- Australia (3):
  - Caboolture
  - Fitzroy
  - Kippa-Ring
- Brazil (3):
  - Curitiba
  - Goiânia
  - São Paulo
- Canada (7):
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Pointe-Claire, Quebec
- Tallinn, Estonia
- Germany (7):
  - Bad Nauheim
  - Berlin
  - Erfurt
  - Erlangen
  - Leipzig
  - München
  - Wiesbaden
- Greece (4):
  - Athens
  - Heraklion
  - Ioannina
  - Thessaloniki
- Dublin, Ireland
- Mexico (4):
  - Guadalajara
  - Mexico City
  - Monterrey
  - San Luis Potosí City
- New Zealand (3):
  - Auckland
  - Christchurch
  - Lower Hutt
- Poland (5):
  - Elblag
  - Sopot
  - Szczecin
  - Torun
  - Warsaw
- South Africa (5):
  - Bloemfontein
  - Cape Town
  - Durban
  - Johannesburg
  - Pretoria
- Spain (7):
  - A Coruña
  - Barcelona
  - Córdoba
  - Lugo
  - Madrid
  - Sabadell
  - San Cristóbal de La Laguna
- United Kingdom (8):
  - Basingstoke
  - Cannock
  - Harrogate
  - Leeds
  - Metropolitan Borough of Wirral
  - Newcastle upon Tyne
  - Southampton
  - Wigan